CLINICAL TRIAL: NCT04623606
Title: Exploratory, Open Label, Multiple Dose, Phase I/II Trial Evaluating Safety, Efficacy of Intravenous and Intraosseous Infusion of Allogeneic Fetal Mesenchymal Stem In Treatment of Severe Osteogenesis Imperfecta Compared With Historical and Untreated Prospective Controls
Brief Title: Boost to Brittle Bones - Stem Cell Transplantation for Treatment of Brittle Bones
Acronym: BOOST2B
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Ministry of Science and Technology, India (Other Government); Vinnova (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Vrisha Madhuri, Professor, Christian Medical College, Vellore, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCB2B0X
Record Dates: First submitted 2020-09-18; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Osteogenesis Imperfecta
Keywords: OI, Brittle bone disease; Hereditary bone fragility
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Intervention Model Description: Historical and Untreated prospective control and Treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Control (Untreated) and historical controls (No Intervention): Subjects eligible for the trial but not willing/able to participate in any of the experimental arms Matched historical controls. Subjects will be identified in historical registries and data will be retrieved from OI database
- Treatment (Experimental): Administration of four doses of BOOST cells with the first dose between 1-4 years of age and the three additional doses at +4, +8 and +12 months after the first dose. Each dose is 3x10^6 MSC/kg body weight.
  Interventions: Biological: BOOST cells

INTERVENTIONS:
Biological: BOOST cells — Four doses of expanded human 1st trimester fetal liver-derived mesenchymal stem cells.
  Arms: Treatment

SUMMARY:
An exploratory, open label, multiple dose, phase I/II trial (n=15) evaluating safety and efficacy of intravenous and intraosseous infusion of allogeneic expanded fetal mesenchymal stem cells (MSC) for the treatment of severe Osteogenesis Imperfecta (OI) compared with historical and untreated prospective controls.

ELIGIBILITY:
(i)Inclusion Criteria Treatment group

1. Parent's/legal guardian's signed informed-consent form
2. Clinical diagnosis of OI type III or IV AND
3. Molecular diagnosis of OI (Glycine substitution in the collagen triple-helix encoding region of either the COL1A1 or COL1A2 gene)
4. Age between 1 to 4 years
5. BP treatment initiated before inclusion
6. Parent/legal guardian over 18 years of age

(ii)Inclusion Criteria Prospective Untreated Control Group and Historical Control Group:

1. Parent's/legal guardian's signed informed-consent form
2. Clinical and molecular diagnosis of OI (Glycine substitution in the collagen triple-helix encoding region of either the COL1A1 or COL1A2 gene)
3. Age between 4 to 8 years
4. Parent/legal guardian over 18 years of age

(iii)Exclusion Criteria Treatment group Prospective and historical control group:

1. Existence of other known disorder that might interfere with the treatment (such as severe malformations, congenital heart defect, hypoxic encephalopathy (l-lll), neurological problems, immune deficiencies, muscle diseases, syndromes) diagnosed by clinical examination
2. Any contraindication for invasive procedures such as a moderate/severe bleeding tendency or contagious infections
3. Abnormal karyotype or other confirmed genetic syndromes
4. Oncologic disease
5. Inability to comply with the trial protocol and evaluation and follow-up schedule
6. Inability to understand the information and to provide informed consent

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability measured as seriousness, severity and frequency of treatment related adverse events (AEs) | From baseline to 16 months follow up
  The primary endpoint is safety and tolerability measured as seriousness, severity and frequency of treatment related adverse events (AEs)/Serious AE (SAE)/Suspected Unexpected Serious Adverse Reaction (SUSAR)with specific focus on the following:
  1. Vital signs in conjunction with the MSC infusion
  2. Transfusion reactions (infusion toxicity, embolism, allergy, infections)
  3. Immune reaction towards the cells, donor-specific antibodies, graft rejection, Graft versus Host Disease, autoimmunity)
  4. Tumourigenicity
  5. Mortality/morbidity

SECONDARY OUTCOMES:
Number of fractures [ Time Frame: From baseline to 16 months follow-up ] | From baseline to 16 months follow up
  Number of fractures.
Time (days) to first fracture after each stem cell administration. [ Time Frame: From each dose of stem cells to the time point of the first fracture. | From baseline to 16 months follow up
  Time (days) to first fracture after each stem cell administration. Number of fractures
Change in bone-marrow density (g/cm2). [ Time Frame: From baseline to the primary follow-up (From baseline to 16 months follow up) | From baseline to 16 months follow up
  Change in bone-marrow density (g/cm2).
Growth (cm). [ Time Frame: From baseline to16 months follow up] | From baseline to 16 months follow up
  Growth (cm) as assessed by clinician
Weight (kg). [ Time Frame: From baseline to 16 months follow up] | From baseline to 16 months follow up
  Growth (kg) as assessed by clinician.
Change in clinical status of OI. [ Time Frame: From baseline to 16 months follow up] | From baseline to 16 months follow up
  Change in clinical status of OI based on parameters defined under efficacy assessments described in protocol, as assessed by OI clinician.
Assessment of biochemical bone turnover by analysis of the markers P-Calcium (mg %) in blood samples. | From at baseline to 16 months follow up
  Assessment of biochemical bone turnover marker P-Calcium (mg %)
Assessment of biochemical bone turnover by analysis of the markers P-Phosphate (mg %) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker P-Phosphate (mg %)
Assessment of biochemical bone turnover by analysis of the markers P-Albumin (g/dL) | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker P-Albumin (g/dL)
Assessment of biochemical bone turnover by analysis of the markers S-ALP (IU/L) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker S-ALP (IU/L)
Assessment of biochemical bone turnover by analysis of the markers S-CTx (mg %) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker S-CTx (mg %)
Assessment of biochemical bone turnover by analysis of the markers fP-PTH (pg/mL)in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker fP-PTH (pg/mL)
Assessment of biochemical bone turnover by analysis of the markers Vitamin D (nmol/L) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker Vitamin D (nmol/L)
Assessment of biochemical bone turnover by analysis of the markers Bone specific S-ALP (μg/L) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker Bone specific S-ALP (μg/L)
Assessment of biochemical bone turnover by analysis of the markers S-Osteocalcin (ng/mL) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker S-Osteocalcin (ng/mL)
Assessment of biochemical bone turnover by analysis of the markers U-DPD/Krea and U-NTx/Krea (mg %) in blood samples. | From baseline to 16 months follow up
  Assessment of biochemical bone turnover marker U-DPD/Krea and U-NTx/Krea (mg %)

OTHER OUTCOMES:
Impact on the subjects Quality of Life: Pediatric Quality of Life Questionnaire™ (PedsQOL) [ Time Frame: From baseline to the 16 month follow-up | From baseline to 16 months follow up
  Quality of life assessed using the Infant Pediatric Quality of Life Questionnaire™ (PedsQOL).
Incidence of donor cells engrafted into patient tissue samples assessed by histology. [ Time Frame: From baseline to the 16 month follow up | From baseline to 16 months follow up
  Donor cell engraftment.
Analysis of an array of cytokines and micro vesicles to evaluate paracrine effects. [ Time Frame: From baseline to the 16 month follow up | From baseline to 16 months follow up
  Paracrine effects will be analysed from plasma isolated from peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Vrisha Madhuri, MS Orth, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No